CLINICAL TRIAL: NCT01311739
Title: An Open-label, Single-Dose, Parallel-Group, Randomized Study of Comparative Bioavailability of B12 After Oral Administration of B2 Formulated With an Absorption Promoter (SNAC), Oral B12 Alone and IV B12 in Healthy Male Subjects
Brief Title: Oral Cyanocobalamin (Eligen B12) Bioavailability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emisphere Technologies, Inc. (Industry)
Responsible Party: M. Cristina Castelli, Ph. D., Emisphere Technologies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMIS 112-C-01
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: Pharmacokinetics
MeSH Terms: interventions — Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10 mg Eligen® B12 (Cyanocobalamin/SNAC) (Experimental): A single oral dose of Eligen® B12, cyanocobalamin/SNAC (5 mg cyanocobalamin/100 mg SNAC) administered in the fasted state as 2 tablets taken with 50 mL of water resulting in a total dose of 10 mg cyanocobalamin and 200 mg SNAC.
  Interventions: Drug: Cyanocobalamin
- 5 mg Eligen® B12 (Cyanocobalamin/SNAC) (Experimental): A single oral dose of Eligen® B12, cyanocobalamin/SNAC (5 mg cyanocobalamin/100 mg SNAC) administered in the fasted state as a tablet taken with 50 mL of water resulting in a total dose of 5 mg cyanocobalamin and 100 mg SNAC.
  Interventions: Drug: Cyanocobalamin
- 5 mg Oral Cyanocobalamin (Active Comparator): A single oral dose of cyanocobalamin alone (5 mg cyanocobalamin, commercial: VITALABS, INC) administered in the fasted state as a tablet taken with 50 mL of water resulting in a total dose of 5 mg cyanocobalamin.
  Interventions: Drug: Cyanocobalamin
- 1 mg Intravenous Cyanocobalamin (Active Comparator): A single intravenous (IV) dose of cyanocobalamin (1 mg cyanocobalamin) administered in the fasted state. Each subject will receive a 1 mL IV injection of a 1 mg/mL (1000 μg/mL) solution resulting in a total dose of 1 mg cyanocobalamin.
  Interventions: Drug: Cyanocobalamin

INTERVENTIONS:
Drug: Cyanocobalamin
  Other Names: B12, Eligen® B12, Cobalamin

SUMMARY:
The purpose of this study is to assess and compare the pharmacokinetics (PK) of cyanocobalamin after the oral administration of Eligen® B12 (cyanocobalamin/SNAC), oral cyanocobalamin alone (commercially-available formulation) and cyanocobalamin administered intravenously (IV) (also a commercially-available formulation) to healthy male subjects under fasting conditions. The safety and tolerability of oral Eligen® B12 (cyanocobalamin/SNAC) versus oral cyanocobalamin alone and versus IV cyanocobalamin are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 45 years.
* Signed ICF prior to any study-related procedures.
* Normal organ function including renal and hepatic function.
* Normal hematological function.
* Body weight between 60 and 100 kg and within 18 - 30 kg/m2 for body mass index (BMI).
* Normal ranges in vital signs, ECG, and laboratory tests.
* Normal ranges of serum B12, methylmalonic acid (MMA), and homocysteine.

Exclusion Criteria:

* Current use (within 14 days) of acetaminophen or non-steroidal anti-inflammatory drugs (NSAIDs) (i.e., aspirin or ibuprofen)
* Current use (within 14 days) of antibiotics, antacids, multivitamins, or nutritional supplements.
* Absolute platelet count below 100 x 109/L
* History or current diagnosis of any clinically significant disease of the liver, kidneys or GI system, or any abnormal condition that compromises the function of these systems and could result in the possibility of altered absorption, excess accumulation, or impairment of metabolism or excretion of the study product.
* History or current diagnosis of any clinically significant hematological, immunological, metabolic, cardiovascular, neurological, or GI abnormalities which that should, in the opinion of the Investigator exclude the subject from this study.
* Any other clinically significant laboratory value at Screening, which, in the opinion of the Investigator, suggested a condition that could have precluded the subject from entering this study.
* At risk of transmitting infection via blood samples e.g., producing a positive HIV test at screening or having participated in a high-risk activity for contracting HIV; producing a positive HBsAg test at screening; producing a positive hepatitis C antibody test at screening.
* Participation in a clinical research study involving a new chemical entity within 30 days of study entry.
* Significant loss or donation of blood within 56 days or plasma within 30 days prior to the initial dose in this study.
* Unsuitable for any reason to receive study product in the opinion of the Investigator.
* Alcohol consumption within the last 48 hours prior to study entry or anytime during the study.
* Positive urine alcohol test.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Serum Cobalamin Pharmacokinetics (PK) | pre-dose to 24 hours post-dose
  Serum cobalamin evaluated via collection and processing of blood samples from predose through 24 hours. Pharmacokinetics to be determined by non-compartmental analysis using predose to 24 hour serum cyanocobalamin non-baseline-adjusted and baseline-adjusted concentration data. Serum cobalamin PK parameters to include: Cmax, tmax, AUClast, AUC∞, t1/2, and Kel and bioavailability (% F) of oral formulations.

SECONDARY OUTCOMES:
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | pre-dose to 24 (end-of-study) hours postdose
  Safety evaluated through the monitoring of medical history findings, physical examination findings, concomitant medications, vital signs (including blood pressure, respiratory rate, heart rate, and temperature), laboratory tests (hematology, serum chemistry, and urinalysis values), ECGs, AEs, and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M. Connolly, MD, Principal Investigator — MDS Pharma Services

REFERENCES:
- [Derived] Castelli MC, Wong DF, Friedman K, Riley MG. Pharmacokinetics of oral cyanocobalamin formulated with sodium N-[8-(2-hydroxybenzoyl)amino]caprylate (SNAC): an open-label, randomized, single-dose, parallel-group study in healthy male subjects. Clin Ther. 2011 Jul;33(7):934-45. doi: 10.1016/j.clinthera.2011.05.088. Epub 2011 Jul 1. PMID 21722960